CLINICAL TRIAL: NCT01819584
Title: Long Term Glucose Metabolism in Conservatively Treated Patients With Congenital Hyperinsulinism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-12-9794-KM-CTIL
Record Dates: First submitted 2013-03-24; First posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Conservatively Treated CHI Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients below 15 years old
- Patients above 15 years old

SUMMARY:
The purpose of this study is to continue follow up of conservatively treated CHI patients and to focus on their metabolic outcome, including frequency of hypoglycemia after discontinuing treatment and incidence of diabetes mellitus in the long term.

ELIGIBILITY:
Inclusion Criteria:

* conservatively treated CHI patients who are in remission for at least one year

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include conservatively treated CHI patients who are in remission for at least one year
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
presence and frequency of hypoglycemia and hyperglycemia. | one year

SECONDARY OUTCOMES:
incidence of diabetes mellitus | 5 years

OTHER OUTCOMES:
presence of metabolic syndrome | 5 years